CLINICAL TRIAL: NCT00391599
Title: Are Enemas Given Before Elective Cesarean Section Useful?
Brief Title: Enemas Before Elective Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Samuel Lurie, Porfessor, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OS-SL-002
Record Dates: First submitted 2006-10-22; First posted 2006-10-24 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-01

CONDITIONS: Complications After Cesarean Section
Keywords: Cesarean Section,; Enema
MeSH Terms: interventions — Enema

ARMS (2):
- Study Group (Experimental): a fleet enema (250 cc of sodium biphosphate 16 gr and sodium phosphate 6 gr per 100 cc) the night before cesarean section
  Interventions: Procedure: enema
- Control Group (Active Comparator): no preoperative intestinal preparation.
  Interventions: Procedure: enema

INTERVENTIONS:
Procedure: enema

SUMMARY:
Enemas are not anymore used routinely before vaginal deliveries.The intention of this study is to elucidate whether there is a benefit in routine use of enema before cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean Section, Elective

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Lurie, MD, Principal Investigator — Edith Wolfson Medical Center

REFERENCES:
- [Derived] Lurie S, Baider C, Glickman H, Golan A, Sadan O. Are enemas given before cesarean section useful? A prospective randomized controlled study. Eur J Obstet Gynecol Reprod Biol. 2012 Jul;163(1):27-9. doi: 10.1016/j.ejogrb.2012.03.034. Epub 2012 Apr 17. PMID 22516178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The inclusion criteria were elective cesarean section and no history of previous abdominal operations except for cesarean delivery.
Groups:
- Study Group: The patients were given a Fleet enema (250 cm3 of sodium biphosphate 16 g and sodium phosphate 6 g/100 cm3) the night before cesarean section
- Control Group: The patients had no preoperative intestinal preparation on the night before cesarean section
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 65 | 65
Completed | 65 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Group: a fleet enema (250 cc of sodium biphosphate 16 gr and sodium phosphate 6 gr per 100 cc) the night before cesarean section
  enema
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (6.1) | 31.3 (5.3) | 31.9 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 65 | 130
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 65 | 65 | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bowel Sounds
Description: bowel sounds: present
Time Frame: On postoperative day 1
Measure: Number; unit: participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 65 | 65
participants | 23 | 31
Statistical Analysis 1: Comparison: Study Group vs Control Group; Test type: Superiority or Other; p = 0.15, Chi-squared

2. Primary Outcome: Number of Participants With Gas Passage
Description: gas passage: present
Time Frame: On postoperative day 1
Measure: Number; unit: participants
Groups:
- Control Group: no preoperative intestinal preparation.
  enema
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 65 | 65
participants | 31 | 34

3. Primary Outcome: Number of Participants Had Spontaneous Feces
Description: occurrence of spontaneous feces
Time Frame: On postoperative day 1
Measure: Number; unit: participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 65 | 65
participants | 1 | 7
Statistical Analysis 1: Comparison: Study Group; Test type: Superiority or Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Groups:
- Study Group: a fleet enema (250 cc of sodium biphosphate 16 gr and sodium phosphate 6 gr per 100 cc) the night before cesarean section
  enema
  the night before cesarean section
- Control Group: no preoperative intestinal preparation.
  the night before cesarean section
Arm/Group | Study Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No